CLINICAL TRIAL: NCT04276025
Title: Relationship Between Histopathological Features, Mutation Status, 18F-FDG PET/CT Radiomic Imaging Parameters as Well as Clinical Outcome in Patients With Treatment-naïve Non-small Cell Lung Cancer
Brief Title: Pathological and Nuclear Medicine Factors for Prognosis in Lung Carcinoma
Acronym: PANU
Status: Completed | Type: Observational
Sponsor: Klinikum Bayreuth GmbH (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Sana Klinikum Hof (Unknown)
Responsible Party: Sponsor
Other Study IDs: PANU022020
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: NSCLC
Keywords: F18-FDG-PET/CT; Radiomics; Texture analysis; Lung cancer; Molecular pathology
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Material from routine diagnosis. No additional material taken from the present study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- German cohort Bayreuth: Retrospective analysis of clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome data.
  Interventions: Other: Clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome
- German cohort Hof: Retrospective analysis of clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome data.
  Interventions: Other: Clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome
- Chinese cohort Beijing: Retrospective analysis of clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome data.
  Interventions: Other: Clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome

INTERVENTIONS:
Other: Clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome — Retrospective analysis of clinical routine F18-FDG-PET/CT, molecular pathology and clinical outcome data.

SUMMARY:
Retrospective study in patients with therapy-naive non small cell lung carcinoma correlating presurgical F18-FDG-PET/CT imaging texture analysis data with postsurgical molecular pathology data and clinical patient outcome. Main aim is to identify pretherapeutic prognostic factors.

DETAILED DESCRIPTION:
Section 1:title and overview Title: Relationship between histopathological features, mutation status, 18F-FDG PET/CT radiomic imaging parameters as well as clinical outcome in patients with treatment-naïve non-small cell lung cancer(NSCLC).

Overview: Nowadays, the most increasingly rapid incidence rate among all tumors is lung cancer, which shows the highest morbidity rate. According to types of tumor cells, lung cancer is divided into two categories: small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC), the latter one includes squamous cell carcinoma, adenocacinoma and large cell carcinoma. The treatment methods are different according to TNM stages, mainly including surgical resection, focal therapy, radiotherapy, chemotherapy as well as immunotherapy. Despite improvements in drug development and treatments for NSCLC patients, five-year survival rates remain unacceptably low, because many patients present with advanced stages at initial diagnosis, with resistancy to therapy and with distant metastases. So an effective way to improve low survival rate is to increase diagnose rate in early stage, to predict whether patients will have benefits from the therapy and to determine probability of distant metastases. Positron emission tomography (PET)/ computed tomography (CT) plays an increasing clinical role in the management of many cancer patients, because it shows additional value in tumor staging, response assessment, prognosis and prediction of treatment response.

Currently, clinical predictive results of PET/CT imaging texture analyses have been obtained in a wide variety of malignancies, such as high-grade gliomas, breast cancer, lung cancer, metastatic colorectal cancer. Most of these studies have shown a significant relationship between PET/CT textural imaging data and patient's clinical outcome. More specifically, a number of NSCLC studies correlated diver gene and a series of PET/CT radiomic imaging parameters, in order to predict clinical outcomes of NSCLC patients.

However the results are somehow controversial and there is no standardization regarding calculation of PET/CT imaging parameters apart from standardized uptake values (SUV). Therefore additional studies are necessary.

Histopathological Lung Cancer Biomarkers:

Lung cancer biomarkers, such as gene mutation, circulating tumor cells (CTCs), have vital effects on predicting pathologic diagnosis, selecting effective therapy decisions and evaluating clinical outcomes accurately. Through the recognitions and utilizing those new biomarkers, the investigators can select the optimal targeted anticancer therapies, and develop new drugs against lung cancer.

Gene biomarkers:

Epidermal growth factor receptor (EGFR) is a tyrosine kinase receptor member of the ERBB family, located on the short arm of chromosome 7 at the position 125. Extracellular ligand binding triggers homodimerization or heterodimerization of ErbB family receptors, phosphorylating active sites in the cytoplasmic tyrosine kinase, and activating intracellular PI3K/AKT/mTOR and RAS/RAF/MAPK pathways. EGFR signaling is critical in development and cellular homeostasis, proliferation, and growth. EGFR and its family members became the important candidates for the development of targeted therapeutics due to the expression rate, 50% in NSCLC, and the relationship between expression rate and poor prognosis.

The B-RAF proto-oncogene, serine/threonine kinase (BRAF) oncogene is located at the long arm of chromosome 7 at position 344. It is involved in the RAS-RAF-MEK-ERK signaling pathway by encoding for a serine/threonine kinase. When activated, BRAF promotes cell growth, proliferation and survival. BRAF was reported mostly in adenocarcinoma and current or former smokers. It has been reported that there are 1%-3% BRAF mutations in NSCLC, and its role as a prognostic predictor.

Anaplastic lymphoma kinase (ALK) is a tyrosine receptor member of the insulin receptor superfamily, locating on the short arm of chromosome 2 at position 2310. And ALK gene rearrangement was described in a subset of NSCLC tumors harboring a fusion of ALK and echinoderm microtubule-associated protein-like 4(EML4) gene. The chimeric protein with constitutive kinase activity encoded by the arrangement promotes malignant growth and proliferation. The EML4-ALK fusion has been detected in 3.7% to 7% of NSCLC and it has a role in prediction of prognosis.

ROS proto-oncogene 1, receptor tyrosine kinase (ROS1) is a tyrosine kinase receptor member of the insulin receptor family and is located on the long arm of chromosome 6 at position 224. It involves in the signal pathways including JAK-ATAT3N, RAS/MEK/ERK, PI3K/AKT and so on. It was reported that about 1% to 2% of NSCLCs harbor ROS1 rearrangements. It occurs in young, female, never smokers with a histologic results of adenocarcinoma. It has a role in prediction.

Recently, an important discovery called "immune checkpoints" has aroused much more attention which means programmed death 1(PD-1) and programmed death-ligand 1 receptor (PD-L1). PD-1, belonging to the CD28 family, is a key immune checkpoint receptor expressing on the surface of the activated T, B and NK cells and plays a crucial role in tumor immune escape. PD-L1 is upregulated in different types of tumors, including NSCLC. PD-L1 delivers negative costimulatory signals and binds PD-1 to reduce cellular immune responses by inducing T-cell apoptosis or exhaustion. Blocking the PD-1/PD-L1 pathway with monoclonal antibodies is currently considered to be the most promising approach, offering durable activity and long-term survival outcomes. The study by Zhang et al. showed that the association between PD-L1 expression and prognosis is dependent on ethnicity. But the role of PD-L1 to predict overall survival is different in studies.

PET/CT Radiomics Imaging Parameters:

Many oncological imaging studies aimed at quantitative assessment of 18F-FDG PET and the correlation with clinical outcomes. There is an underling hypothesis on which radiomics glucose metabolism parameters rely on the existence of a relationship between extracted metabolic image data and tumor molecular phenotype and/or genotype. Radiomic parameters ideally may determine patient prognosis and predict clinical patient outcomes, being divided into two types of parameters: A) conventional PET/CT parameters and B) textural features.

Conventional PET/CT parameters include different basic metabolic parameters and volumetric parameters , such as SUVMAX, SUVMEAN, SUVPEAK, MTV, TLG, which are more or less routinely obtained and many times used in clinical patients reports.

Textural PET/CT features represent more advanced metabolic parameters and are currently not in clinical use. They are considered to demonstrate i.e. the spatial heterogeneity of malignant tumors including second-order parameters, high-order, such as GLCM, GLRLM, and GLSZM. Such advanced textural PET/CT features seem to perform better than the conventional PET/CT parameters used for imaging explanation in clinical routine. However, to date there is no consensus considering optimal segmentation methods or quantitative indices to express metabolic characteristics of a tumor leision and which textural PET/CT features can be used for clinical diagnostic purposes. Therefore, more standardized studies are needed to conclude an optimal method and to allow those parameters to be used in clinical routine diagnostics in cancer patients.

Section 2：purpose and method

Purpose:

1. to select those PET/CT radiomic imaging parameters which are most robust and repeatable after evaluation with two different published calculation methods and cross-validate using two different patient collectives (German and chinese NSCLC patients);
2. to evaluate the relationship between the type of gene mutations, conventional and textural PET/CT parameters and clinical outcomes in patients with treatment-naïve NSCLC;
3. to evaluate the relationship between CTCs, conventional and textural PET/CT parameters and clinical outcome in patients with treatment-naïve NSCLC.

Method： PET/CT radiomic imaging parameters calculation: perform post-proccessing of quality assessed, reconstructed, attenuation corrected 18F-FDG PET images and obtain conventional 18F-FDG PET/CT parameters SUVMAX, SUVMEAN, SUVPEAK, TLG, MTV using the "MM Oncology" application within the SIEMENS Syngo.via Software. Obtain textural PET/CT features, using two different previously published softwares, LIFEx and MATLAB script, to extract all textural parameters. Then compare the results of the textural parameters obtained with two different softwares and select which ones are most robust and repeatable considering the differently acquired methods. Determine which textural parameters show the same changing trends in order to remove redundant ones.

The investigators will cooperate with two well known departments (Nuclear Medicine and Pathology) specialized in oncology (Peking University Cancer Hospital) sharing anonymized patient data in NSCLC patients, in order to expand sample size, to cross-validate data and to compare similarities and differences between patients regarding different races and different regions as well as different imaging analysis methods in order to make the main results more reliable. After establishment and validation of this two-site-platform the plan is to expand analyses examining additional solid tumors such as malignant melanoma etc.

The investigators plan to extract proteins expressed by mutant genes from CTCs and analyze which gene mutations are determined. To determine the correlation between genetic mutations identified in CTCs and gene mutations identified by histopathological biopsy.

Section 3: advantage and limitation Advantage: as far as known, this is the first multisite study examining a German and a Chinese NSCLC patient collective using the same scan protocol on the same PET/CT scanner, examining different published software programs to extract and calculate 18F-FDG PET/CT textural features, making our results more understandable and more reliable and offering a possibility to cross-validate our analyses.

Limitation：the retrospective character of the study, which will not allow us to draw any definite conclusions regarding parameter selection for clinical routine purposes.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective selection of both German cohort NSCLC patients with concomitant gene mutation results, CTCs accounting results and 18F-FDG PET/CT imaging data before lung tumor surgery (both German patient cohorts)
* Retrsopective selection of Chinese NSCLC patients with concomitant gene mutation results, CTCs accounting results and 18F-FDG PET/CT imaging data before lung tumor surgery (Chinese patient collective)

Exclusion Criteria:

* NSCLC patients with surgical resection of the target/primary tumor before 18F-FDG PET/CT scanning.
* NSCLC patients with elevated blood glucose levels (> 150 mg/dl) immediately before 18F-FDG injection.
* based on PET CT scanning no concomitant malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German and chinese NSCLC patients who have received presurgical F18-FDG-PET/CT imaging followed by surgical removal of the primary lung tumor with postsurgical molecular pathology evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | through study completion an average of 3 years after initial inclusion
  Time to progression (RECIST) based on routine clinical CT imaging on a quarterly base
Overall survival | through study completion an average of 3 years after initial inclusion
  Time to death based on clinical records

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu QG, Zhang SM, Ding XX, He B, Zhang HQ. Driver genes in non-small cell lung cancer: Characteristics, detection methods, and targeted therapies. Oncotarget. 2017 Apr 10;8(34):57680-57692. doi: 10.18632/oncotarget.17016. eCollection 2017 Aug 22. PMID 28915704
- [Background] O'Flaherty L, Wikman H, Pantel K. Biology and clinical significance of circulating tumor cell subpopulations in lung cancer. Transl Lung Cancer Res. 2017 Aug;6(4):431-443. doi: 10.21037/tlcr.2017.07.03. PMID 28904887
- [Background] Sollini M, Cozzi L, Antunovic L, Chiti A, Kirienko M. PET Radiomics in NSCLC: state of the art and a proposal for harmonization of methodology. Sci Rep. 2017 Mar 23;7(1):358. doi: 10.1038/s41598-017-00426-y. PMID 28336974
- [Background] Villalobos P, Wistuba II. Lung Cancer Biomarkers. Hematol Oncol Clin North Am. 2017 Feb;31(1):13-29. doi: 10.1016/j.hoc.2016.08.006. PMID 27912828
- [Background] Khalil FK, Altiok S. Advances in EGFR as a Predictive Marker in Lung Adenocarcinoma. Cancer Control. 2015 Apr;22(2):193-9. doi: 10.1177/107327481502200210. PMID 26068764
- [Background] Sholl LM. Biomarkers in lung adenocarcinoma: a decade of progress. Arch Pathol Lab Med. 2015 Apr;139(4):469-80. doi: 10.5858/arpa.2014-0128-RA. Epub 2014 Sep 25. PMID 25255293
- [Background] Sharma SV, Bell DW, Settleman J, Haber DA. Epidermal growth factor receptor mutations in lung cancer. Nat Rev Cancer. 2007 Mar;7(3):169-81. doi: 10.1038/nrc2088. PMID 17318210
- [Background] Cardarella S, Ogino A, Nishino M, Butaney M, Shen J, Lydon C, Yeap BY, Sholl LM, Johnson BE, Janne PA. Clinical, pathologic, and biologic features associated with BRAF mutations in non-small cell lung cancer. Clin Cancer Res. 2013 Aug 15;19(16):4532-40. doi: 10.1158/1078-0432.CCR-13-0657. Epub 2013 Jul 5. PMID 23833300
- [Background] Paik PK, Arcila ME, Fara M, Sima CS, Miller VA, Kris MG, Ladanyi M, Riely GJ. Clinical characteristics of patients with lung adenocarcinomas harboring BRAF mutations. J Clin Oncol. 2011 May 20;29(15):2046-51. doi: 10.1200/JCO.2010.33.1280. Epub 2011 Apr 11. PMID 21483012
- [Background] Zhao Z, Verma V, Zhang M. Anaplastic lymphoma kinase: Role in cancer and therapy perspective. Cancer Biol Ther. 2015;16(12):1691-701. doi: 10.1080/15384047.2015.1095407. PMID 26529396
- [Background] Fujimoto J, Wistuba II. Current concepts on the molecular pathology of non-small cell lung carcinoma. Semin Diagn Pathol. 2014 Jul;31(4):306-13. doi: 10.1053/j.semdp.2014.06.008. Epub 2014 Jun 12. PMID 25239274
- [Background] Chatziandreou I, Tsioli P, Sakellariou S, Mourkioti I, Giannopoulou I, Levidou G, Korkolopoulou P, Patsouris E, Saetta AA. Comprehensive Molecular Analysis of NSCLC; Clinicopathological Associations. PLoS One. 2015 Jul 24;10(7):e0133859. doi: 10.1371/journal.pone.0133859. eCollection 2015. PMID 26208325
- [Background] Yoshida A, Kohno T, Tsuta K, Wakai S, Arai Y, Shimada Y, Asamura H, Furuta K, Shibata T, Tsuda H. ROS1-rearranged lung cancer: a clinicopathologic and molecular study of 15 surgical cases. Am J Surg Pathol. 2013 Apr;37(4):554-62. doi: 10.1097/PAS.0b013e3182758fe6. PMID 23426121
- [Background] Intlekofer AM, Thompson CB. At the bench: preclinical rationale for CTLA-4 and PD-1 blockade as cancer immunotherapy. J Leukoc Biol. 2013 Jul;94(1):25-39. doi: 10.1189/jlb.1212621. Epub 2013 Apr 26. PMID 23625198
- [Background] Zou W, Wolchok JD, Chen L. PD-L1 (B7-H1) and PD-1 pathway blockade for cancer therapy: Mechanisms, response biomarkers, and combinations. Sci Transl Med. 2016 Mar 2;8(328):328rv4. doi: 10.1126/scitranslmed.aad7118. PMID 26936508
- [Background] Ameratunga M, Asadi K, Lin X, Walkiewicz M, Murone C, Knight S, Mitchell P, Boutros P, John T. PD-L1 and Tumor Infiltrating Lymphocytes as Prognostic Markers in Resected NSCLC. PLoS One. 2016 Apr 22;11(4):e0153954. doi: 10.1371/journal.pone.0153954. eCollection 2016. PMID 27104612
- [Background] Ma W, Gilligan BM, Yuan J, Li T. Current status and perspectives in translational biomarker research for PD-1/PD-L1 immune checkpoint blockade therapy. J Hematol Oncol. 2016 May 27;9(1):47. doi: 10.1186/s13045-016-0277-y. PMID 27234522
- [Background] Zhang M, Li G, Wang Y, Wang Y, Zhao S, Haihong P, Zhao H, Wang Y. PD-L1 expression in lung cancer and its correlation with driver mutations: a meta-analysis. Sci Rep. 2017 Aug 31;7(1):10255. doi: 10.1038/s41598-017-10925-7. PMID 28860576
- [Background] Pan ZK, Ye F, Wu X, An HX, Wu JX. Clinicopathological and prognostic significance of programmed cell death ligand1 (PD-L1) expression in patients with non-small cell lung cancer: a meta-analysis. J Thorac Dis. 2015 Mar;7(3):462-70. doi: 10.3978/j.issn.2072-1439.2015.02.13. PMID 25922726
- [Background] Zhong A, Xing Y, Pan X, Shi M, Xu H. Prognostic value of programmed cell death-ligand 1 expression in patients with non-small-cell lung cancer: evidence from an updated meta-analysis. Onco Targets Ther. 2015 Dec 1;8:3595-601. doi: 10.2147/OTT.S91469. eCollection 2015. PMID 26664143
- [Background] van Helden EJ, Vacher YJL, van Wieringen WN, van Velden FHP, Verheul HMW, Hoekstra OS, Boellaard R, Menke-van der Houven van Oordt CW. Radiomics analysis of pre-treatment [18F]FDG PET/CT for patients with metastatic colorectal cancer undergoing palliative systemic treatment. Eur J Nucl Med Mol Imaging. 2018 Dec;45(13):2307-2317. doi: 10.1007/s00259-018-4100-6. Epub 2018 Aug 9. PMID 30094460
- [Background] Cook GJR, Azad G, Owczarczyk K, Siddique M, Goh V. Challenges and Promises of PET Radiomics. Int J Radiat Oncol Biol Phys. 2018 Nov 15;102(4):1083-1089. doi: 10.1016/j.ijrobp.2017.12.268. Epub 2018 Jan 31. PMID 29395627
- [Background] Chicklore S, Goh V, Siddique M, Roy A, Marsden PK, Cook GJ. Quantifying tumour heterogeneity in 18F-FDG PET/CT imaging by texture analysis. Eur J Nucl Med Mol Imaging. 2013 Jan;40(1):133-40. doi: 10.1007/s00259-012-2247-0. Epub 2012 Oct 13. PMID 23064544
- [Background] Pyka T, Gempt J, Hiob D, Ringel F, Schlegel J, Bette S, Wester HJ, Meyer B, Forster S. Textural analysis of pre-therapeutic [18F]-FET-PET and its correlation with tumor grade and patient survival in high-grade gliomas. Eur J Nucl Med Mol Imaging. 2016 Jan;43(1):133-141. doi: 10.1007/s00259-015-3140-4. Epub 2015 Jul 29. PMID 26219871
- [Background] Nioche C, Orlhac F, Boughdad S, Reuze S, Goya-Outi J, Robert C, Pellot-Barakat C, Soussan M, Frouin F, Buvat I. LIFEx: A Freeware for Radiomic Feature Calculation in Multimodality Imaging to Accelerate Advances in the Characterization of Tumor Heterogeneity. Cancer Res. 2018 Aug 15;78(16):4786-4789. doi: 10.1158/0008-5472.CAN-18-0125. Epub 2018 Jun 29. PMID 29959149
- [Background] Orlhac F, Soussan M, Maisonobe JA, Garcia CA, Vanderlinden B, Buvat I. Tumor texture analysis in 18F-FDG PET: relationships between texture parameters, histogram indices, standardized uptake values, metabolic volumes, and total lesion glycolysis. J Nucl Med. 2014 Mar;55(3):414-22. doi: 10.2967/jnumed.113.129858. Epub 2014 Feb 18. PMID 24549286
- [Result] Pyka T, Bundschuh RA, Andratschke N, Mayer B, Specht HM, Papp L, Zsoter N, Essler M. Textural features in pre-treatment [F18]-FDG-PET/CT are correlated with risk of local recurrence and disease-specific survival in early stage NSCLC patients receiving primary stereotactic radiation therapy. Radiat Oncol. 2015 Apr 22;10:100. doi: 10.1186/s13014-015-0407-7. PMID 25900186